CLINICAL TRIAL: NCT01214395
Title: An Investigator Blinded Controlled Study of the Nasal Application of 5% Tea Tree Oil (TTO) for the Prevention of Catheter-associated Infections in Renal Dialysis Patients
Brief Title: Nasal Tea Tree Oil for the Prevention of Infections in PD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PathWest Laboratory Medicine WA (Other Government)
Responsible Party: Principal Investigator, Kerry Carson, Co-Investigator, PathWest Laboratory Medicine WA
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006-199
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: haemodialysis; peritoneal dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 5% tea tree oil nasal ointment — daily for 5 days then weekly for 6 months

SUMMARY:
This study will compare the use of tea tree oil as a topical nasal antiseptic to prevent infections in patients that need renal dialysis. A maximum of fifty subjects will be recruited and will be assessed for signs of infection once per week for the first 6 weeks and then every 4 weeks until week 26. They will also be checked for nasal carriage of 'Golden Staph' when they enroll in the trial. The subjects will complete the trial if they have 26 weeks infection-free or if they have an infection during that period

DETAILED DESCRIPTION:
The patients for the trial are to be recruited in the Renal Unit at SCGH and at enrolment a nasal swab is taken to see if the patients has nasal carriage of S. aureus. The patient is also given a prescription for 5% TTO nasal ointment which was filled by the SCGH pharmacy. The application of medication will follow the usual procedure which consists of bi-daily nasal application for 5 days and then weekly application for the next 25 weeks of the trial. The patients are not blinded and are given all their medication at one dispensing which consists of 3 × 10 g tubes of 5% TTO. The patients have weekly assessments for the first 6 weeks of the trial and then 4 weekly assessments until week 26. All assessments are conducted during routine dressing changes or routine visits and are conducted by specially trained dialysis nurses. During each visit the catheter site is examined for any signs of infection and the findings documented on a questionnaire. Suspected cases of infection are identified by trained nurses and the consultant physician will then examined the patient. The findings will be documented by the nurse on a questionnaire and submitted to the primary investigator for review, confirmation, and classification. The primary endpoint is the proportion of patients with a catheter-related infection within 6 months after entry into the study. The infections included: (1) exit site infection (ESI); (2) tunnel infections; and (3) bacteraemia. The endpoint is evaluated by the primary investigator according to the definitions for catheter-related infections. Cases with "definite" and "probable" infections will be classified as infections.

All catheter-related infections are treated by the patient's nephrologist according to their usual practice. If a new catheter is clinically indicated, the patient will continued to receive the same ointment to which they had been assigned. Swabs for cultures and sensitivities at the catheter exit site are taken if an exit or tunnel infection is suspected and blood cultures if a bacteraemia is suspected. All microbiology samples will be sent to the PathWest laboratory for culture and sensitivities. The study will end when the last enrolled subject has completed the minimum 6-month study period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age
* A signed and dated written informed consent is obtained prior to participation.
* Able to comply with the requirements of the protocol.
* Have ESRD and dialysis is planned
* Requirement either haemodialysis or peritoneal dialysis

Exclusion Criteria:

* known sensitivity to TTO
* Use of mediated and non-medicated nasal ointments in the past 12 weeks
* HD patients likely to transfer to a another dialysis centre in the next 6 months
* Re-insertion of CVC
* serious, uncontrolled disease (including serious psychological disorders) likely to interfere with the study and/or likely to cause death within the study duration
* participation in another clinical trial during the last 12 weeks
* previous participation in this trial
* known contraindication to any component of mupirocin
* concurrent diseases which exclude the administration of therapy as outlined by the study protocol
* active infections requiring systemically administered antibiotics or antiviral medications within the last 7 days
* acute renal failure
* non-compensated heart failure
* myocardial infarction during the last 6 months
* chronic lung disease with hypoxemia
* severe non-compensated hypertension
* severe non-compensated diabetes mellitus
* known HIV or active chronic hepatitis B or C infection
* subjects who, in the opinion of the investigator, are not likely to complete the study for what ever reason.
* subjects who, in the opinion of the investigator, abuse alcohol or drugs
* subjects with any clinically significant abnormality (to be determined by the investigator) following review of screening laboratory data and full physical examination. Stable medical conditions unlikely to affect patient safety or the outcome of the investigation may be acceptable if agreed by the study monitor appointed by the sponsor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hutchison, MBBS, Principal Investigator — Sir Charles Gairdner Hospital
Locations (1):
- Sir Charles Gairdner Hospital, Perth, Western Australia, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from the Renal Unit at Sir Charles Gairdner Hospital and was conducted by the nursing staff in that ward. The recruitment period was from 1 July 2010-30 June 2011.
Pre-assignment Details: All enrolled patients participated in the trial.
Groups:
- Tea Tree Oil Application: tea tree oil medication group
Period: Overall Study
Arm/Group | Tea Tree Oil Application
Started | 5
Completed | 0
Not Completed | 5
Not completed — All patients had infection | 5

BASELINE CHARACTERISTICS:
Arm/Group | Tea Tree Oil Application
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  Australia | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint Will be the Number of Tea Tree Oil Patients That Did Not Have a Catheter-related Infection Within 6 Months After Entry Into the Trial.
Description: Catheter-related infections will be defined according to standard guidelines
  Cases with "definite" and "probable" infections will be classified as infections.
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Tea Tree Oil: tea tree oil application
Arm/Group | Tea Tree Oil
Number analyzed (Participants) | 5
participants | 0

2. Secondary Outcome: The Number of Patients That Did Not Have a Staphylococcus Aureus Infection
Time Frame: 6 months
Population: counted
Measure: Number; unit: participants
Groups:
- Did Not Have Staph. Aureus Infection: No exit site infection or peritonitis with Staph. aureus
Arm/Group | Did Not Have Staph. Aureus Infection
Number analyzed (Participants) | 5
participants | 3

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Tea Tree Oil Application
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tea Tree Oil Application (N=5)
peritonitis (Renal and urinary disorders) | 2 (2) — Hospitalisation for peritonitis. Two patients were hospitalised - one with an infection and the other for metabolic peritonitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No